CLINICAL TRIAL: NCT01914614
Title: A Pilot Study of Working Women and Breast Cancer
Status: Completed | Type: Observational
Sponsor: Robin Vanderpool (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Robin Vanderpool, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: IRB # 13-0560-P3H; K12DA035150 (NIH)
Record Dates: First submitted 2013-07-26; First posted 2013-08-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Working Women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Working Poor Survivors: Low Wage workers
- Non-Working Poor Survivors: Higher-Wage Salary Workers

SUMMARY:
The purpose of this research is to better understand the relationship between employment and breast cancer. Research is being conducted to understand how workplace factors influence breast cancer patients' ability to adhere to recommended cancer treatment and effectively recover from cancer. Investigators hope to use the findings from the study to help working breast cancer survivors make informed decisions about treatment and employment in collaboration with their employers and healthcare providers.

DETAILED DESCRIPTION:
Patients enrolled will be interviewed three times over a six month period. They will be asked questions about their experiences in managing their cancer while taking care of their job responsibilities. Patients will be asked to complete a survey that asks questions about their breast cancer treatment, their job, and how they manage their responsibilities while undergoing cancer treatment.

The first initial meeting will be conducted at a time and location that is convenient for the patient. This meeting should last about an hour to an hour and a half.

Three and six months after the initial interview, study participants will be asked to complete a follow-up survey by either telephone or Internet/Web, depending on their preference. These telephone surveys will last between 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-65
* Working at least 20 hours per week
* Currently patients of the University of Kentucky Markey Cancer Center
* Are able to read, write, and communicate in English
* Have reliable telephone or Internet/Web access in or outside the home

Exclusion Criteria:

* Self-employed
* Unemployed
* Cognitively impaired

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with a new, primary breast cancer within 3 months of enrollment and who were employed at the time of diagnosis.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Guideline concordant breast cancer treatment as defined by National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology and oncologist assessments. | 6 months
  Differences in receipt of guideline-concordant breast cancer treatment between working poor and working non-poor survivors as explained by variations in occupation and work organization factors associated with each group of women. Guideline-concordant treatment will be informed by National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology and oncologist assessments.

SECONDARY OUTCOMES:
Breast cancer treatment adherence, including completion of prescribed chemotherapy regimens, prescribed radiation treatment regimen, and/or surgical follow-up appointments. | 6 months
  Differences in breast cancer treatment adherence rates between working poor and non-poor survivors as explained by variations in occupation and work organization factors associated with each group of women.
Satisfaction with breast cancer treatment decision-making | 6 months
  Differences in satisfaction with breast cancer treatment decision-making between working poor and working non-poor survivors as explained by variations in occupation and work organization factors associated with each group of women.
Quality of life | 6 months
  Differences in quality of life measures between working poor and working non-poor survivors explained by variations in occupation and work organization factors associated with each group of women.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Vanderpool, DrPH, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Center for Clinical and Translational Science, Lexington, Kentucky
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky